CLINICAL TRIAL: NCT01334606
Title: Evaluation of Glycemic Control and User Acceptability of the BD Ultra-Fine Nano 4 mm x 32G Pen Needle for Injection of Long-acting or Basal Insulin Doses Above 40 Units
Brief Title: Evaluation of a 4mmx32G Pen Needle for Injection of Basal Insulin Doses Above 40 Units
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated due to unanticipated recruitment difficulties.
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DBC-10-SQUIR04
Record Dates: First submitted 2011-04-08; First posted 2011-04-13 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; pen needle; basal insulin; long-acting insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nano: 4mm x 32G Pen Needle (Experimental): Subjects will use the 4mm x 32G pen needle for all self-administered pen injections of diabetes medications during the assigned three week study period.
  Interventions: Device: 4 mm x 32G pen needle (Nano)
- Short: 8mm x 31G Pen Needle (Experimental): Subjects will use the 8 mm x 31G pen needle for all self-administered pen injections of diabetes medications during the assigned three week study period.
  Interventions: Device: 8mm x 31G pen needle (Short)

INTERVENTIONS:
Device: 4 mm x 32G pen needle (Nano) — The pen needle will be used to administer all pen-based diabetes medications. When using the 4mm Nano pen needle, subjects are directed to hold the pen device at a 90 degree angle and perform the injection with no pinch-up.
  Other Names: 4 mm x 32 G BD Ultra-Fine Nano pen needle
  Arms: Nano: 4mm x 32G Pen Needle
Device: 8mm x 31G pen needle (Short) — The pen needle will be used to administer all pen-based diabetes medications. When using the 8mm Short pen needle, subjects are directed to use the pinch-up technique for injections in the abdomen and thigh, and no pinch-up at other injection sites. Subjects are to hold the pen device at a 90 degree angle.
  Other Names: 8 mm x 31G BD Ultra-Fine Short insulin pen needle.
  Arms: Short: 8mm x 31G Pen Needle

SUMMARY:
The primary purpose of this study is to demonstrate that the BD 4mm x 32G Ultra-Fine Nano pen needle provides equivalent glycemic control to the BD 8mm x 31G Ultra-Fine short pen needle as measured by fructosamine (FRU) among Lantus®, Levemir®, and/or NPH users taking one or more single daily injections of greater than 40 units of insulin.

Glycemic control, injection pain, leakage, preference, comfort, and other parameters will be compared between the 4mm x 32G and the 8 mm x 31 G pen needle after three weeks of use of each device. Sufficient numbers of subjects taking Lantus® as their basal insulin will be enrolled so as to allow for pre-specified analysis of this subgroup.

DETAILED DESCRIPTION:
This is an open-label, randomized two period crossover study. Each subject's participation is expected to last about seven weeks and includes a brief enrolment period followed by two consecutive three week treatment periods (Period 1 and Period 2).

In Period 1, subjects will use the first assigned study pen needle (either the 4mm Nano or the 8mm Short) to self-administer daily all their pen-based diabetes medications. Upon completion of Period 1, subjects will switch to the alternate pen needle for Period 2. The randomization schedule will determine the order of pen needle use.

Blood samples for determination of fasting blood glucose and serum fructosamine concentrations will be collected at baseline (Visit 2) and the end of Period 1 (Visit 3) and Period 2 (Visit 4). Blood samples will be analyzed by a central laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus
* Have been using a pen device for all diabetes or diabetes-related medications for at least one month prior to screening
* Use a pen device to self-administer greater than 40 units of Lantus, Levemir, and/or NPH in one or more single injections. For split doses, at least one of the injections must deliver more than 40 units.
* Documented hemoglobin A1c (HbA1c) from 5.5% to 9.5%, inclusive
* Self monitor blood glucose at once daily with a memory blood glucose meter, and willing do so at least twice per day for the duration of the study
* On a stable diabetes regimen (insulin and non-insulin meds, diet and exercise) for at least 1 month prior to screening
* Able to read, write and follow instructions in English

Exclusion Criteria:

* Current administration of insulin with a pump.
* Current use a syringe to inject insulin or any diabetes-related medication
* Participation in clinical study BDDC-08-011 or DBC-10-SQUIR05
* History of intravenous drug abuse.
* Current status or history of a medical condition that would contraindicate treatment with study products or other conditions which, in the opinion of the Investigator, would place the subject at risk or potentially confound interpretation of the study results (i.e., recent history of ketoacidosis, hypoglycemic unawareness, etc).
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence J Hirsch, MD, Study Director — BD Medical - Diabetes Care
Locations (3):
- United States (2):
  - International Diabetes Center (IDC), Minneapolis, Minnesota
  - Comprehensive Clinical Research, Berlin, New Jersey
- BioPharma Services Inc., Toronto, Ontario, Canada

REFERENCES:
- [Background] Hirsch LJ, Gibney MA, Li L, Berube J. Glycemic control, reported pain and leakage with a 4 mm x 32 G pen needle in obese and non-obese adults with diabetes: a post hoc analysis. Curr Med Res Opin. 2012 Aug;28(8):1305-11. doi: 10.1185/03007995.2012.709181. Epub 2012 Jul 18. PMID 22762347
- [Background] Hirsch LJ, Gibney MA, Albanese J, Qu S, Kassler-Taub K, Klaff LJ, Bailey TS. Comparative glycemic control, safety and patient ratings for a new 4 mm x 32G insulin pen needle in adults with diabetes. Curr Med Res Opin. 2010 Jun;26(6):1531-41. doi: 10.1185/03007995.2010.482499. PMID 20429832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began at three medical research centers in March 2011. Due to slow enrolment, the study was terminated after 9 weeks.
Pre-assignment Details: There is no information for this section.
Groups:
- All Study Participants: Since only 3 subjects completed both periods of the crossover study before it was prematurely terminated, the primary endpoint analysis could not be performed. Therefore, no tabulations by intervention were prepared.
Period: Overall Study
Arm/Group | All Study Participants
Started | 21
Completed | 3
Not Completed | 18
Not completed — Study Terminated due to slow enrolment | 18

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This includes all subjects randomized to either intervention sequence. Since only 3 subjects completed both study periods, the data are not presented by intervention.
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 16
  Canada | 5

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control as Measured by Percent (%) Absolute Change in Fructosamine
Description: The measure of glycemic control will be the percent difference in FRU assessed at the end of Period 1 compared to FRU assessed at the end of Period 2. The average percent difference in FRU between the Nano and Short pen needles, with the Short as a reference, must be shown to be no more than +/- 20% with 95% confidence. General linear models will be used, adjusting for baseline FRU. This outcome measure was to be determined for the total subject population as well as for the subset of Lantus users.
Time Frame: 3 weeks per pen needle
Population: No analysis was performed. The study was terminated due to slow enrollment. The same endpoint was studied and reported in a similar subject population, including Lantus users, in study DBC-11-SQUIR05(NCT01231984)which had a similar design.
Groups:
- All Subjects: Due to early termination of the study, only 3 subjects completed both study periods. Analysis of the primary outcome measure requires FRU data from both study periods. Due to the lack of sufficient data, no analysis was performed.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the start of study participation until subjects completed, or were discontinued from the study. Subjects that participated in the study used each pen needle for up to 3 weeks.
Groups:
- All Study Participants: This includes all subjects that participated in the study. A total of 22 adverse events were reported. The investigator reported that 14 of 22 events were not related to the study product, and 8 of 22 events were unlikely related to the study product.
- 4mmx32G Pen Needle: Subjects that used the 4mmx32G pen needle, either during Study Period 1 or Study Period 2
- 8mmx31G Pen Needle: Subjects that used the 8mmx31G pen needle, either during Study Period 1 or Study Period 2
Arm/Group | All Study Participants | 4mmx32G Pen Needle | 8mmx31G Pen Needle
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/21 | 0/21
Other Adverse Events (participants affected / at risk) | 9/21 | 6/21 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=21) | 4mmx32G Pen Needle (N=21) | 8mmx31G Pen Needle (N=21)
Progressive Degeneration right knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) — Hospitalized for total right knee arthroplasty. Not related to study participation.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=21) | 4mmx32G Pen Needle (N=21) | 8mmx31G Pen Needle (N=21)
Tennis Elbow (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
hypoglycemia (Endocrine disorders) | 6 (15) | 3 (3) | 5 (12)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less